CLINICAL TRIAL: NCT02366052
Title: Nutritional Counseling Versus Nutritional Supplements for the Treatment of NASH - a Randomized Prospective, Open Label Pilot Study (Nuces NASH)
Brief Title: Nutritional Counseling vs. Nutritional Supplements for NASH - a Randomized Prospective, Open Label Pilot Study
Acronym: NucesNASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: University of Jena (Other)
Responsible Party: Principal Investigator, Priv.-Doz. Dr. J. Schattenberg, Attending Physician, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUCES_NASH-JGU; SCHA 1015/5-1 (Other Grant/Funding Number: DFG)
Record Dates: First submitted 2013-11-01; First posted 2015-02-19 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Non-alcoholic Fatty Liver Disease; Fatty Liver, Nonalcoholic
Keywords: Histologically confirmed NASH; Hepatocyte Injury determined by M30 antigen
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nutritional Counseling (Active Comparator): The nutritional counseling group will receive dietary counseling focusing on a reduction of fructose intake by a trained nutritionist for 12 weeks every 3 weeks.
  Interventions: Behavioral: Nutritional Counseling
- Nutritional Counseling and LCS (Experimental): The dietary supplement LCS (Lactobacillus casei shirota ) will be given 2 times a day for 12 weeks in addition to the nutritional counseling every 3 weeks.
  Interventions: Other: Nutritional Counseling and LCS
- Lactobacillus Casei Shirota (Experimental): The dietary supplement LCS (Lactobacillus casei shirota ) will be given 2 times a day for 12 weeks.
  Interventions: Dietary Supplement: Lactobacillus casei shirota (LCS)

INTERVENTIONS:
Behavioral: Nutritional Counseling — Nutritional counseling by a trained nutritionist for 12 weeks.
  Arms: Nutritional Counseling
Dietary Supplement: Lactobacillus casei shirota (LCS) — The dietary supplement LCS (Yakult plus) will be given 2 times a day for 12 weeks in addition to dietary counseling every 3 weeks.
  Other Names: Yakult plus
  Arms: Lactobacillus Casei Shirota
Other: Nutritional Counseling and LCS — Nutritional counseling by a trained nutritionist in addition to the dietary supplement LCS (2 times a day) for 12 weeks.
  Other Names: Nutritional Counseling and Yakult plus
  Arms: Nutritional Counseling and LCS

SUMMARY:
The main aim of the study is to determine if an oral supplementation of the LCS has a beneficial effect by itself or even enhances the beneficial effects of a moderate life-style intervention on the progression of NAFLD in humans.

ELIGIBILITY:
Inclusion Criteria:

- Elevated M30 antigen levels (cutoff: >200 - 800 U/L) at screening AND hepatic steatosis on ultrasound

OR histologically confirmed NASH

- Age 18 to 75 years

Exclusion Criteria:

* Alcohol intake of more than 30 g/d (men) or 20 g/d (women)
* Treatment with ursodeoxycholic acid (UDCA), Vitamin E or other investigational NASH drugs 3 months prior to randomization
* Treatment with medications or substances that may induce secondary NASH (e.g., tamoxifen, corticosteroids, amiodarone, methotrexate) or ameliorate NASH (TNF-antagonists)
* Treatment with phenprocoumon or warfarin
* Hepatocellular carcinoma or non-hepatic malignancy
* Decompensated cirrhosis (Child B,C) or a history of decompensation
* Liver disease unrelated to NASH, including chronic viral hepatitis B/D or C, autoimmune hepatitis, Wilson's disease or clinical manifest iron overload
* Bariatric surgery within the last 5 years
* BMI <18,5 kg/m2 or BMI >45 kg/m2
* Liver transplantation
* Heart failure (New York Heart Association Class II - IV)
* Myocardial infarction, instable coronary artery disease , coronary artery intervention or stroke in the previous 6 months
* Instable chronic obstructive pulmonary disease, chronic inflammatory bowel disease or rheumatoid arthritis.
* Instable renal insufficiency (changes in serum creatinin > 50% in the last 3 month) or terminal renal insufficiency requiring dialysis
* Uncontrolled hypertension (blood pressure > 180/90 despite therapy)
* Uncontrolled diabetes mellitus defined by hemoglobin A1c > 9
* Food allergies requiring strictly dietary adherence
* Pregnant or nursing women
* Chronic pancreatitis or history of recurring acute pancreatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Reduction of the M30 antigen in the serum | 12 and 24 weeks
  Reduction of the M30 antigen as a validated measure of the degree of hepatocellular inflammation and injury

SECONDARY OUTCOMES:
Change in indicators of hepatocellular injury and fibrosis | 12 and 24 weeks
  Change in indicators of hepatocellular injury (ALT, gammaGT, M30/M60 antigen ratio, ELF score), proinflammatory cytokines (hsCRP, ferritin, plasminogen activator-1, endotoxin), surrogate parameters of liver fibrosis (fibrosis marker panels, Fibrotest, ELF score) and relative liver stiffness (assessed by Fibro Scan)
Change in metabolic risk factors | 12 and 24 weeks
  Changes in metabolic risk factors (BMI, waist circumference, Homeostasis Model Assessment/Matsuda Score, serum lipids), changes in oral glucose tolerance and changes in hepatic steatosis will be assessed.
Saftey and tolerability | 12 and 24 weeks
  Safety is assessed by (1) clinical examination, (2) clinical chemistries including serum electrolytes, renal, liver function tests and markers of pancreatic injury.

OTHER OUTCOMES:
Improvement in measures of nutritional physiology | 12 and 24 weeks
  Improvement of nutritional physiology, compliance, self-perceived efficacy, emotional eating behavior using a validated questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jörn M Schattenberg, MD, Principal Investigator — Johannes Gutenberg Universität; Ina Bergheim, PhD, Principal Investigator — Universität Jena
Locations (2):
- Germany (2):
  - Institut für Ernährungswissenschaften, University Jena, Jena
  - University Medical Center of the Johannes Gutenber Univeristy, Mainz